CLINICAL TRIAL: NCT04635124
Title: Optimal Dog Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Optimal dog visits
Record Dates: First submitted 2020-11-16; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Dementia; Aging
Keywords: Animal-assisted therapy; visiting dog; non-pharmacological; nursing home
MeSH Terms: conditions — Dementia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The design of the study is a stratified and randomized complete block design. Each nursing home is a block. The participants are allocated randomly to one of the three visit types (1) Visits with a dog, no activity (D); 2) Visits with a dog, with activity (DA); or 3) Visits without dog, with an activity (A), balancing for the level of cognitive impairment, measured by the MMSE-scale. This was achieved by ranking the participants according to MMSE score within sex and allocating them to the three visit types by using different numerical orders in each nursing home (1, 2, 3; 3, 1, 2; 2, 3, 1 etc.).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1: Dog visit with a dog, no additional activity (D) (Active Comparator): The nursing home resident receives 12 10-minute visits in their own room. The visitor is accompanied with a dog, and the resident can touch the dog. Apart from the visitor, an observer is present.
  Interventions: Behavioral: Dog visit
- 2: Dog visit with an additional activity (DA) (Experimental): The nursing home resident receives 12 10-minute visits in their own room. The visitor is accompanied with a dog, and the resident can touch the dog. During the visit, the visitor offers the resident to participate in an activity that involves interacting with the dog.
  Apart from the visitor, an observer is present.
  Interventions: Behavioral: Dog visit; Behavioral: Encourage to engage in activity
- 3: Visit without dog, with an additional activity (A) (Active Comparator): The nursing home resident receives 12 10-minute visits in their own room. During the visit, the visitor offers the resident to participate in an activity.
  Apart from the visitor, an observer is present, but no dog is present..
  Interventions: Behavioral: Encourage to engage in activity

INTERVENTIONS:
Behavioral: Dog visit — An visitor visits the participant with a dog
  Arms: 1: Dog visit with a dog, no additional activity (D); 2: Dog visit with an additional activity (DA)
Behavioral: Encourage to engage in activity — In each visit the visitor invites the participant to engage in an activitty
  Arms: 2: Dog visit with an additional activity (DA); 3: Visit without dog, with an additional activity (A)

SUMMARY:
The aim of this project is to study how an the intensity of dog contact during dog visits in nursing homes can affect the immediate response to, and the general effect of the visits, and whether the residents' level of cognitive impairment affects the response and benefit of dog visits.

The participants are randomly assigned to receive one type of visits (12 visits in total) out of three possible visit types (1: visit with a dog; 2: visit with a dog, including a planned activity, 3 visit without a dog, including a planned activity). The residents received 2 visits per week for 6 weeks. The behaviour of the participants during visits is recorded. Before and after the intervention period, participants are scores on psychometric scales for cognitive impairment level, daily function level and symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

• Being able to sit up during the visits

Exclusion Criteria:

* Dog allergy
* Fear of dogs
* Health problems that make participation unadvisable

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Behavioural response during visits | Behaviour is recorded in all of the 12 visits in the 6 week intervention period
  The behaviour of the residents is recorded by direct observation using continuous recording. In all visits, the frequency and duration of talk and physical contact to the persons present are recorded. Talk is classified into talk about the dog and/or activity, depending on the visit type. In visits with dogs (D, DA), the frequency and duration of physical contact and talk directed to the dog are recorded, and in visits involving an activity (DA, A), the frequency and duration of the residents' involvement in the activity are recorded.

SECONDARY OUTCOMES:
Cognitive impairment level, before intervention | This measure is obtained in the week preceeding the intervention period (6 weeks, 2 visits )
  All participants were scored on the Mini-Mental State Examination (MMSE), which gives information about the participants' cognitive status.The MMSE score has a minimum and maximum value of 0 and 30, respectively. The lower the score, the more severe the cognitively impairment level.
Daily function level, before intervention | This measure is obtained in the week preceeding the intervention period (6 weeks, 2 visits )
  All participants were scored on The Gottfries-Bråne-Steen Scale (GBS), which is an evaluation of disabilities, language, psychiatric symptoms, average daily living function, and behaviour of the participants. The GBS score has a minimum and maximum value of 0 and 156, respectively. The lower the score, the more well-functioning the patient.
Symptoms of depression, before intervention | This measure is obtained in the week preceeding the intervention period (6 weeks, 2 visits )
  All participants were scored on the Geriatric Depression Scale (GDS), to screen for symptoms of depression. The GDS score has a minimum and maximum value of 0 and 15, respectively.A high score indicates more symptoms of depression.
Cognitive impairment level, after intervention | This measure is obtained in the week following the intervention period (6 weeks, 2 visits )
  All participants were scored on the Mini-Mental State Examination (MMSE), which gives information about the participants' cognitive status. The MMSE score has a minimum and maximum value of 0 and 30, respectively. The lower the score, the more severe the cognitively impairment level.
Daily function level,, after intervention | This measure is obtained in the week following the intervention period (6 weeks, 2 visits )
  All participants were scored on The Gottfries-Bråne-Steen Scale (GBS), which is an evaluation of disabilities, language, psychiatric symptoms, average daily living function, and behaviour of the participants. The GBS score has a minimum and maximum value of 0 and 156, respectively. The lower the score, the more well-functioning the patient.
Symptoms of depression, after intervention | This measure is obtained in the week following the intervention period (6 weeks, 2 visits )
  All participants were scored on the Geriatric Depression Scale (GDS), to screen for symptoms of depression. The GDS score has a minimum and maximum value of 0 and 15, respectively.A high score indicates more symptoms of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Thodberg, Principal Investigator — University of Aarhus

IPD SHARING:
Plan to Share IPD: No